CLINICAL TRIAL: NCT06727591
Title: Evaluation of Horizontal Anterior Mandibular Augmentation With Split Bone Block Technique From the Chin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: hossam samy mohamed saleh (Other)
Responsible Party: Sponsor-Investigator, hossam samy mohamed saleh, Principal Investigator, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #8/2023
Record Dates: First submitted 2024-12-04; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Alveolar Bone Grafting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Horizontal Ridge Augmentation with Split Bone Block (Experimental)
  Interventions: Procedure: Split Bone Block Technique

INTERVENTIONS:
Procedure: Split Bone Block Technique — An intraoral crestal incision with/out vertical arms was performed on alveolar ridge using blade no.15. After flap reflection, patroning the defect to help guide the area to be grafted from the donor site. At the chin area (donor site) unicortical cuts will be made at least 5 mm inferior to root tips, 5 mm superior to inferior border of mandible and 5 mm away from the mental foramen. The graft was luxated and split into two bone shells each 1 ~ 2 mm in thickness using disc. The bone shells and the donor site were scrapped for autogenous graft particles. Decortication of the recipient site. The graft was stabilised into the recipient site using two or more self tapping titanium screws placed midway corono-apical in the bone shell following the ridge contour. The autogenous particles were packed into the space between the split bone block and the ridge. Collagen sponge was used to cover the donor site. After 4 months the site was approached for implant placement using crestal incision

SUMMARY:
The aim of this study was to compare clinically and radiographically bone gain, healing of the surgical site, healing of the grafted bone and stability of the grafted area following horizontal ridge augmentation at anterior mandible using split bone block from the chin area.

ELIGIBILITY:
Inclusion Criteria:

* Patient with missing anterior mandibular teeth
* horizontal bone width < 5 mm
* Adequate zone of keratinized tissue

Exclusion Criteria:

* Presence of infection or periapical lesions in adjacent teeth
* Medically compromised patients with a condition that affect the procedure
* Insufficient inter-arch distance
* Bruxism or clenching
* Alcoholism
* Smokers

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | up to 2 weeks
  It was assessed through a 10-point Visual Analogue Scale (VAS). The categories were as follows (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe)
Implant stability | up to 3 months
  Implant stability was measured using Osstell. Osstell measures the resonance frequency which indicated the implant stability. It has a scale from 1 to 100 where:
  * <60 is considered low stability.
  * 60 ~ 69 is considered intermediate stability.
  * ≥ 70 is considered high stability
Amount of horizontal bone gain | up to 4 months
  This was measured on cone beam computed tomography (CBCT) by comparing pre- and post-operative bone width at specific levels around the implant.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt